CLINICAL TRIAL: NCT06934434
Title: Evaluation of Familial Mediterranean Fever (FMF) Impact on Oral and Dental Health in Children and Adolescents
Brief Title: Evaluation of Familial Mediterranean Fever Impact on Oral and Dental Health in Children and Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ozge Gungor (Other)
Collaborators: Akdeniz University (Other)
Responsible Party: Sponsor-Investigator, Ozge Gungor, pHd, DDS, Assoc. Prof. Dr. Pediatric Dentist, Akdeniz University
Organization: Akdeniz University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: AkdenizUıremkapıcı002
Record Dates: First submitted 2025-04-09; First posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: FMF
Keywords: FMF; DMFT; Saliva; bruxism; Oral health
MeSH Terms: conditions — Bruxism | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study group with FMF (Experimental): The study group was named 'Study group with FMF'.
  Interventions: Other: FMF Study Group
- Healthy control group (Experimental): The control group consisting of healthy participants was called 'Healthy control group'.
  Interventions: Other: control group

INTERVENTIONS:
Other: FMF Study Group — In the study group consisting of children with FMF, DMFT, dft, bruxism, tooth wear due to bruxism, gingival index (MGI), plaque index (OHI-S), salivary pH, salivary flow rate, salivary buffering capacity, dental age, chronological age difference, mesio-distal dimensions of the teeth, and the presence of aphthous lesions were determined.
  Arms: Study group with FMF
Other: control group — In the control group consisting of healthy children, DMFT, dft, bruxism, tooth wear due to bruxism, gingival index (MGI), plaque index (OHI-S), salivary pH, salivary flow rate, salivary buffering capacity, dental age, chronological age difference, mesio-distal dimensions of the teeth, and the presence of aphthous lesions were determined.
  Arms: Healthy control group

SUMMARY:
Aim: It is the clinical and radiological evaluation of oral hygiene, teeth and surrounding tissues in children and adolescents diagnosed with FMF and comparing the results with healthy individuals. Method: Our study included patients aged 6-15, 45 with FMF (study group) and 45 healthy (control group), who were referred from Akdeniz University Faculty of Medicine Pediatric Rheumatology Clinic and evaluated at Akdeniz University Faculty of Dentistry Pedodontics Clinic. MEFV gene mutations were investigated in the study group. After recording the demographic and clinical characteristics of both groups, intraoral examinations were performed and DMFT, dft, bruxism, tooth wear due to bruxism and gingival/plaque indexes were evaluated. Saliva pH, flow rate and buffering capacity were measured. Tooth age was determined by the Cameriere method, The mesio-distal dimensions of the teeth were measured on the plaster model.

DETAILED DESCRIPTION:
In the study, DMFT, dft, bruxism, tooth wear due to bruxism, gingival index (MGI), plaque index (OHI-S), salivary pH, salivary flow rate, salivary buffering capacity, dental age, chronological age difference, mesio-distal dimensions of the teeth, and the presence of aphthous lesions were evaluated and compared between the study group consisting of children with FMF and the control group of healthy children.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with FMF, aged between 6-15 years, who were admitted/referred to the Pediatric Dentistry Department Clinic of Akdeniz University Faculty of Dentistry for oral and dental examination, and who agreed to participate in the study after being thoroughly informed both verbally and in writing.
* Patients with no systemic diseases other than FMF.
* Patients who have not used any systemic antibiotics or similar medications (e.g., antidepressants, psychiatric drugs) within the last 3 months.

Exclusion Criteria:

* Patients diagnosed with FMF, who were admitted/referred to the Pediatric Dentistry Department Clinic of Akdeniz University Faculty of Dentistry for oral-dental examination but declined to participate in the study after being thoroughly informed both verbally and in writing.
* Patients with any systemic disease other than FMF.
* Patients who have used systemic antibiotics or any other medications (e.g., antidepressants, psychiatric drugs) within the last 3 months.

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2021-02-05 (Actual); Primary Completion 2021-05-18 (Actual); Study Completion 2022-03-22 (Actual)

PRIMARY OUTCOMES:
DMFT index | 3 months
  To determine the DMFT index score, decayed teeth in permanent teeth are indicated as "D", lost teeth extracted due to decay are indicated as "M", and filled teeth are indicated as "F". The DMFT index is calculated by adding the D, M, F values and dividing them by the total number of permanent teeth. An increase in the calculated scores indicates that oral and dental health is negatively affected.
dft index | 3 months
  The dft Index is the calculated form of the DMFT index for primary teeth. When calculating the dft group index, missing teeth are not included in the calculation. Because it is difficult to diagnose the reason for the loss of primary teeth and there is a high probability of error. For this reason, the number of decayed and filled teeth is calculated during the examination. Decayed teeth are indicated with "d" and filled teeth with "f". The dft index is calculated by adding the d and f values and dividing them by the total number of permanent teeth. An increase in the calculated scores indicates that oral and dental health is negatively affected
Saliva pH | 3 months
  Salivary pH was measured using pH indicator strips. A low pH (<6.5) indicates an acidic environment and increases the risk of tooth demineralization and caries, whereas a high pH (>7.5) indicates an alkaline state, which may be linked to decreased bacterial activity but may also indicate systemic conditions.
Unstimulated salivary flow rate | 3 months
  Unstimulated salivary flow rate is measured by collecting unstimulated saliva over a period of time and calculating the volume per minute. A low flow rate (<0.1 mL/min) indicates hyposalivation, which increases the risk of caries and oral infection, while a high flow rate may be associated with conditions such as gastroesophageal reflux or medication effects.
Saliva buffering capacity | 3 months
  Saliva buffering capacity was measured using the GC Saliva Buffer Kit, which uses a scoring system based on color changes. A low buffering capacity indicates a higher risk of dental caries and enamel demineralization, whereas a high buffering capacity indicates better protection against acid attacks in the oral environment.
Simplified Oral Hygiene Index (OHI-S) | 3 months
  The Simplified Oral Hygiene Index (OHI-S) assesses oral cleanliness by measuring debris and calculus accumulation on selected tooth surfaces. Higher scores indicate poorer oral hygiene, while lower scores suggest better maintenance.
The Modified Gingival Index (MGI) | 3 months
  The Modified Gingival Index (MGI) evaluates gingival inflammation without probing, based on visual inspection. Higher scores reflect increased inflammation and potential periodontal issues.

CONTACTS AND LOCATIONS:
Overall Officials: Özge GÜNGÖR, PhD, DDS, Assoc. Prof. Dr., Principal Investigator — Akdeniz University
Locations (1):
- Akdeniz University Faculty of Dentistry, Department of Pediatric Dentistry,, Antalya, Konyaaltı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No